CLINICAL TRIAL: NCT06590714
Title: Perioperative Polmacoxib Reduce Opioid Consumption for Post Operative Pain After Rotator Cuff Tear.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eulji University Hospital (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Man Kwak, Assistant Professor of Orthopedics, Eulji University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEMC 2024-06-015
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; reduction of Opioids; Effects of Polmacoxib Administration
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Rotator cuff tear patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental(Acelex cap 2mg) (Experimental): Experimental Arm (Polmacoxib (Acelex cap 2mg) + Non-NSAID Non-Opioid or Opioid Analgesics(ULTRACET ER SEMI TAB))
  1. Polmacoxib (preventive Acelex cap 2mg) administration, Method: One tablet orally once daily, regardless of meals.
  Interventions: Drug: Experimental(Acelex cap m2mg)
- Active Comparator(NSAIDs-excluded non-opioid or opioid analgesics) (Active Comparator): Control Group (Administration of Non-NSAID Non-Opioid or Opioid Analgesics(ULTRACET ER SEMI TAB))
  1. Non-NSAID Non-Opioid or Opioid Analgesics(ULTRACET ER SEMI TAB), Administration Method: PRN
  Interventions: Drug: Active Comparator(NSAIDs-excluded non-opioid or opioid analgesics)

INTERVENTIONS:
Drug: Experimental(Acelex cap m2mg) — Experimental Arm (Polmacoxib (Acelex cap 2mg + NSAIDs-excluded non-opioid or opioid analgesics))
  Polmacoxib (preventive Acelex cap 2mg) administered, dosage: 1 tablet orally once daily, regardless of meals.
  NSAIDs-excluded non-opioid or opioid analgesics, dosage: as needed (PRN).
  Arms: Experimental(Acelex cap 2mg)
Drug: Active Comparator(NSAIDs-excluded non-opioid or opioid analgesics) — NSAIDs-excluded non-opioid or opioid analgesics, dosage: as needed (PRN).
  Arms: Active Comparator(NSAIDs-excluded non-opioid or opioid analgesics)

SUMMARY:
1. **One day (±1 day) before surgery:** The investigator or designated study staff will thoroughly explain the clinical trial process to the participant and their guardian (representative) based on the informed consent form and provide the form so that all participants and their guardians have sufficient time to read, discuss, and decide. Participants who agree to participate in the clinical trial will voluntarily sign the written consent form and receive a copy of the signed consent form before any study-related procedures are conducted. The clinical trial site will assign a screening number to patients who voluntarily provide consent and undergo screening. The screening number can be assigned in the order in which the participants sign the consent within the study site. After confirming eligibility based on inclusion/exclusion criteria, randomization will be performed to assign participants to either the treatment group or the control group (with a 1:1 ratio). If assigned to the treatment group, participants will receive 'Polacoxib (preventive Acelex cap 2mg) once daily, NSAIDs-excluded non-opioid/opioid analgesics - PRN use.' If assigned to the control group, participants will receive NSAIDs-excluded non-opioid or opioid analgesics. Data will be collected by comparing the two groups in a double-arm setup. Pain scores, UCLA/ASES scores, and joint range of motion will be collected, and this data will be valid up to 3 months before the surgery. (For patients taking NSAIDs or Ultracet, the dose will be maintained until v5.)
2. **Two hours before surgery:** Administration of medication begins.
3. **Three days after surgery:** Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses (post-surgery). Non-opioid or opioid analgesics (e.g., Fentanyl injection or Ultracet) will be used to manage post-surgical pain, and the number of doses will be collected to assess the participant's pain.
4. **Two weeks after surgery:** An outpatient visit will be conducted one week after discharge. Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses at the two-week mark.
5. **Six weeks after surgery:** Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses.
6. **Three months after surgery:** MRI will be performed to check for re-tears (optional for participants). This visit will be the study's completion visit, during which pain scores, UCLA/ASES scores, joint range of motion, and cumulative doses of NSAIDs-excluded non-opioid or opioid analgesics will be collected. If adverse events occurring during the treatment period have resolved before this completion visit, no additional safety follow-up will be performed, and this visit will be considered the end of the clinical trial. If adverse events have not resolved by the completion visit, follow-up will continue until the adverse events have either returned to pre-study or baseline levels, or the principal investigator or designee determines that the adverse events have stabilized, or no further follow-up is deemed necessary. This follow-up will mark the completion of the clinical trial.

DETAILED DESCRIPTION:
**⑧-1. Visit 0: Pre-surgery Admission, Orthopedic Ward (Consent Acquisition and Screening)** According to the investigator's judgment, patients who are considered potential candidates will be encouraged to participate in the clinical trial. One day (±1 day) before surgery, the investigator or designated study staff will thoroughly explain the clinical trial process to the participant and their guardian (representative) based on the informed consent form and provide the form so that all participants and their guardians have sufficient time to read, discuss, and decide. Participants who agree to participate in the clinical trial will voluntarily sign the written consent form and receive a copy of the signed consent form before any study-related procedures are conducted. The clinical trial site will assign a screening number to patients who voluntarily provide consent and undergo screening. The screening number can be assigned in the order in which the participants sign the consent within the study site. After confirming eligibility based on inclusion/exclusion criteria, randomization will be performed to assign participants to either the treatment group or the control group (with a 1:1 ratio). If assigned to the treatment group, participants will receive 'Polmacoxib (preventive Acelex cap 2mg) once daily,' and NSAIDs-excluded non-opioid/opioid analgesics - PRN. If assigned to the control group, participants will receive NSAIDs-excluded non-opioid or opioid analgesics. Data will be collected by comparing the two groups in a double-arm setup. Pain scores, UCLA/ASES scores, and joint range of motion will be collected, and this data will be valid up to 3 months before the surgery.

**Visit 0 Investigations and Examinations:**

1. Obtain written consent
2. Assign screening number
3. Verify inclusion/exclusion criteria
4. Collect baseline information of the participant
5. Collect baseline disease information
6. Physical examination
7. Imaging data (MRI, X-ray, etc.)
8. UCLA/ASES scores (including pain scores)
9. Joint range of motion
10. Randomization

    * 2. Visit 1: Two Hours Before Surgery, Orthopedic Ward (Medication Administration)** Medication administration begins two hours before surgery.

**Visit 1 Investigations and Examinations:**

1. Medication administration

   * 3. Visit 2: Post-surgery Admission, Orthopedic Ward (Three Days After Surgery)** Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses (post-surgery) three days after surgery. Non-opioid or opioid analgesics (e.g., Fentanyl injection or Ultracet) will be used to manage post-surgical pain, and the number of doses will be collected to assess the participant's pain.

**Visit 2 Investigations and Examinations:**

1. Pain scores
2. Physical examination
3. Check for adverse events
4. Cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses (post-surgery)

   * 4. Visit 3: Two Weeks After Surgery (±3 Days), Orthopedic Outpatient Clinic** An outpatient visit will be conducted one week after discharge. Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses at the two-week mark.

**Visit 3 Investigations and Examinations:**

1. Pain scores
2. Physical examination
3. Check for adverse events
4. Cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses (cumulative since surgery)

   * 5. Visit 4: Six Weeks After Surgery (±3 Days)** Collect pain scores and the cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses at the six-week mark.

**Visit 4 Investigations and Examinations:**

1. Pain scores
2. Cumulative number of NSAIDs-excluded non-opioid or opioid analgesic doses (cumulative since surgery)
3. Physical examination
4. Check for adverse events

   * 6. Visit 5: Twelve Weeks After Surgery (±3 Days), Orthopedic Outpatient Clinic** An MRI will be performed to check for re-tears (optional for participants). This visit will be the study's completion visit, during which pain scores, UCLA/ASES scores, joint range of motion, and cumulative doses of NSAIDs-excluded non-opioid or opioid analgesics will be collected. If adverse events occurring during the treatment period have resolved before this completion visit, no additional safety follow-up will be performed, and this visit will be considered the end of the clinical trial. If adverse events have not resolved by the completion visit, follow-up will continue until the adverse events have either returned to pre-study or baseline levels, or the principal investigator or designee determines that the adverse events have stabilized, or no further follow-up is deemed necessary. This follow-up will mark the completion of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* Patients who need rotator cuff rupture or rotator cuff surgery with MRI identified osteoarthritis (especially small and medium SST dominant rupture)
* NSAIDs unadministered patients for more than 1 month
* Ultracet unadministered patients for more than 1 month

Exclusion Criteria:

* primary fiftieth shoulder
* including short-lived frozen shoulders
* infectious arthritis
* previous corticosteroid injections/surgery
* moderate-severe arthroplasty
* a traumatized patient
* a central or peripheral nervous system disease
* a mental illness that may not conform to medical or physical therapy
* a woman of childbearing age
* Pregnancy
* a severe gastrointestinal ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure-Cumulative administration frequency of narcotic analgesics (e.g., Fentanyl injection), excluding NSAIDs | At postoperative day 3
  Postoperative pain in subjects is managed during the hospital stay by administering non-narcotic or narcotic analgesics, excluding NSAIDs (e.g., Fentanyl injection). Pain levels are assessed by collecting data on the frequency of administration.

SECONDARY OUTCOMES:
Secondary Outcome Measure-Cumulative number of doses of non-opioid analgesics excluding NSAIDs | - 3 days post-surgery - 2 weeks post-surgery - 6 weeks post-surgery - 12 weeks post-surgery
  - Cumulative number of doses of non-opioid analgesics excluding NSAIDs (e.g., Ultracet)
Secondary Outcome Measure-Range of Motion (ROM) | 1 day before surgery, 12 weeks post-surgery
  Range of Motion (ROM)
Secondary Outcome Measure-Rotator cuff re-tear status | 12 weeks post-surgery
  Rotator cuff re-tear status
Secondary Outcome Measure | - 1 day before surgery - 2 weeks post-surgery - 6 weeks post-surgery - 12 weeks post-surgery
  * VAS pain scale
  * The VAS pain scale can be expressed using 11 levels, represented by numbers from 0 to 10. In this case, the patient selects a number that corresponds to the intensity of the pain they are experiencing, ranging from 0 (no pain) to 10 (the worst imaginable pain).
  The meaning of each number is as follows:
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-9: Severe pain 10: Worst possible pain
Primary Outcome Measure-ASES score | 1 day before surgery, 12 weeks post-surgery
  * ASES Score
  * The ASES Score (American Shoulder and Elbow Surgeons Score) is a standardized tool used to assess shoulder function and pain. It provides an objective measurement of shoulder conditions and treatment outcomes by evaluating both subjective pain and functional status.
  The ASES score consists of two key components:
  Pain Assessment: Patients rate their pain intensity on a numeric scale from 0 to 10, where 0 means no pain and 10 indicates severe pain.
  Functional Assessment: It includes 10 questions that evaluate daily shoulder and arm function. Each question is scored from 0 to 3, and this component plays a crucial role in assessing the patient's ability to perform daily activities.
  The final ASES score is calculated on a scale of 0 to 100, with higher scores indicating better shoulder function and less pain. This score helps healthcare professionals monitor shoulder conditions and evaluate treatment effectiveness.
Secondary Outcome Measure-UCLA score | 1 day before surgery, 12 weeks post-surgery
  * UCLA Score
  * The UCLA Shoulder Rating Scale is a standardized tool used to assess shoulder function and pain. It is commonly utilized to evaluate postoperative outcomes or to diagnose shoulder-related conditions.
  The UCLA score is based on five components, totaling a maximum of 35 points:
  Pain (10 points): Evaluates the intensity of the patient's pain. Function (10 points): Assesses the patient's ability to use the shoulder in daily activities.
  Range of Motion (5 points): Measures the range of motion in the shoulder. Strength (5 points): Assesses the strength of the shoulder and arm. Patient Satisfaction (5 points): Evaluates how satisfied the patient is with their shoulder condition.
  Score Interpretation:
  34-35 points: Excellent 28-33 points: Good 21-27 points: Fair 20 points or below: Poor The UCLA score provides a comprehensive assessment of shoulder pain and function, making it particularly useful for tracking recovery after procedures like arthroscopic shoul

CONTACTS AND LOCATIONS:
Locations (1):
- Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24043481/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16762702/